CLINICAL TRIAL: NCT05299138
Title: Restoring Empowerment and Choosing Hope (REACH) in Sarasota Florida
Brief Title: Restoring Empowerment and Choosing Hope (REACH)
Acronym: REACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish Family & Children's Service of the Suncoast, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20220208
Record Dates: First submitted 2022-03-03; First posted 2022-03-28 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Intervention; Wait List Control
Keywords: Healthy relationships, economic self-sufficiency
MeSH Terms: interventions — Marriage; Methods

STUDY DESIGN:
Intervention Model Description: The Intervention group will start with assigning a Case Manager and begin Marriage and Relationship Enhancement Skills (MRES) class weekly and meet with their Case Manager as needed.
Who Masked: Outcomes Assessor
Masking Description: The outside evaluators will remain blind to each condition throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Marriage and Relationship Enhancement Skills (MRES) Intervention (Experimental): The Intervention group will be assigned a Case Manager and begin Marriage and Relationship Enhancement Skills (MRES) class weekly and meet with their Case Manager as needed.
  Interventions: Behavioral: Marriage and Relationship Enhancement Skills (MRES) Intervention
- Wait list control (No Intervention): The Control group will be placed on a wait-list and offered services as soon as they complete the study's final 22-week follow-up measures. Control participants will not be assigned a Case Manager and will not receive any comparable services from our agency until they complete their 22-week measures.

INTERVENTIONS:
Behavioral: Marriage and Relationship Enhancement Skills (MRES) Intervention — The Intervention group will be assigned a Case Manager and placed in the next available Marriage and Relationship Enhancement Skills (MRES) class that is convenient for their schedule. Intervention participants will attend classes weekly and meet with their Case Manager weekly, bi-weekly, or monthly, as needed. Study measures will be gathered from intervention participants at baseline, 10 weeks after baseline, and then 22 weeks after baseline. The following tools will be utilized at baseline and follow-up assessment: (1) REACH program eligibility screening (only conducted at baseline), (2) Information, Family Outcomes, Reporting, and Management (nFORM) system, (3) Family Environment Scale (FES), (4) Revised Dyadic Adjustment Scale (RDAS), and (5) Economic Self-Sufficiency Scale (ESS).
  Arms: Marriage and Relationship Enhancement Skills (MRES) Intervention

SUMMARY:
The goals of REACH are to help adults develop the skills they need to develop healthy relationship and marriage skills, improve ability to parent and co-parent effectively, identify and enhance skills and abilities required to gain or retain economic self-sufficiency, and foster family stability and increase successful marriage rates. Data from the tri-county region comprised of Sarasota, Manatee, and Charlotte counties demonstrates the presence of a number of risk factors affecting family stability, including high rates of single-parent households, births to unwed mothers, and high median rent costs compared to poverty rates and income. By providing families with relationship enhancement, parenting, and economic self-sufficiency services, this should help to optimize each family member's quality of life and improve child well-being.

DETAILED DESCRIPTION:
REACH will serve a minimum of 337 individual adults during each full year of the five-year grant term in Sarasota, Manatee, and Charlotte counties on the Gulf Coast of Florida. REACH will target individual participants and, in cases where both members of a couple are interested in participating, will deliver services to each partner individually. The primary target population for REACH is low-income, at-risk individuals.

Coupled with its successful history of providing healthy marriage programming, JFCS is well-positioned to help families in crisis become more stable and self-sufficient. Understanding the inextricable link between financial security and family stability, REACH is targeting and reaching the most vulnerable individuals based solely on economic risk factors. REACH will incorporate a comprehensive employment program combining both job and career advancement. This will help families in crisis reach improved financial stability, which will in turn improve the ability of individual participants to be better parents and better partners, furthering the goal of promoting healthy marriages and reducing local divorce rates.

ELIGIBILITY:
Inclusion Criteria:

* adults age 18 or older
* interested in education about strengthening their current marriage or committed relationship
* reside in Sarasota, Manatee, and Charlotte counties on the Gulf Coast of Florida

Exclusion Criteria:

* under age 18
* do not reside in Sarasota, Manatee, and Charlotte counties

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Family Environment Survey (FES) | 22 weeks after baseline
  The FES was developed to measure social and environmental characteristics of families. Face and content validity are supported by clear statements about family situations that relate to subscale domains, and the measure can differentiate between distressed and normal family samples.

SECONDARY OUTCOMES:
Revised Dyadic Adjustment Scale (RDAS) | 22 weeks after baseline
  The RDAS is a 32-item self-report standardized measure with 4 subscales (Dyadic Consensus, Dyadic Satisfaction, Affectional Expression, Dyadic Cohesion) in addition to a total score.

OTHER OUTCOMES:
Economic Self-Sufficiency Scale (ESS) | 22 weeks after baseline
  The ESS includes the following subscales with demonstrated reliability and validity: 1) Financial Management Attitudes Scale, 2) Scale of Economic Self-Sufficiency, 3) Financial Knowledge Scale, 4) Family Empowerment Scale, and 5) Financial Management and Planning Behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Katelyn Kopakin, MA, Study Director — Jewish Family Children's Services of the Suncoast, Inc.
Locations (1):
- Jewish Family and Children Service, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: No